CLINICAL TRIAL: NCT01126736
Title: An Open-Label, Multicenter, Randomized Phase Ib/II Study of Eribulin Mesylate Administered in Combination With Pemetrexed Versus Pemetrexed Alone as Second Line Therapy in Patients With Stage IIIB or IV Nonsquamous Non Small Cell Lung Cancer
Brief Title: Eribulin Mesylate Administered in Combination With Pemetrexed Versus Pemetrexed Alone as Second Line Therapy in Patients With Stage IIIB or IV Nonsquamous Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-701; 2009-016047-19 (EudraCT Number)
Record Dates: First submitted 2010-05-17; First posted 2010-05-20 (Estimated); Results first posted 2022-08-04 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: neoplams; lung neoplasms; Stage IIIB; IV Nonsquamous Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — eribulin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose E7389 in Combination with Pemetrexed (Experimental)
  Interventions: Drug: eribulin mesylate
- Pemetrexed (Active Comparator)
  Interventions: Drug: pemetrexed
- High Dose E7389 in Cominbation with Pemetrexed (Experimental): Eribulin mesylate (eribulin; E7389) administered as a 2-5 minute intravenous (IV) bolus in one of two dosing schedules for both the Phase Ib and Phase 2 portions: either Days 1 and 8 of a 21 day cycle in ascending doses of 0.7, 1.1, or 1.4 mg/m2 or on Day 1 of the 21-day cycle at doses at ascending doses of 0.9, 1.4, or 2.0 mg/m2.
  Interventions: Drug: Eribulin mesylate (eribulin; E7389)

INTERVENTIONS:
Drug: eribulin mesylate — Eribulin mesylate (eribulin; E7389) administered as a 2-5 minute intravenous (IV) bolus in one of two dosing schedules for both the Phase Ib and Phase 2 portions: either Days 1 and 8 of a 21 day cycle in ascending doses of 0.7, 1.1, or 1.4 mg/m2 or on Day 1 of the 21-day cycle at doses at ascending doses of 0.9, 1.4, or 2.0 mg/m2.
  Other Names: halichrondrin B analog; Alimta
  Arms: Low Dose E7389 in Combination with Pemetrexed
Drug: pemetrexed — Pemetrexed given at a dose of 500 mg/m2 as an IV infusion on Day 1 of a 21-day cycle. Patients will also receive dexamethasone and vitamin supplements as recommended in the prescribing information for pemetrexed.
  Other Names: halichrondrin B analog; Alimta
  Arms: Pemetrexed
Drug: Eribulin mesylate (eribulin; E7389) — Eribulin mesylate (eribulin; E7389) administered as a 2-5 minute intravenous (IV) bolus in one of two dosing schedules for both the Phase Ib and Phase 2 portions: either Days 1 and 8 of a 21 day cycle in ascending doses of 0.7, 1.1, or 1.4 mg/m2 or on Day 1 of the 21-day cycle at doses at ascending doses of 0.9, 1.4, or 2.0 mg/m2.
  Arms: High Dose E7389 in Cominbation with Pemetrexed

SUMMARY:
The purpose of this study is to determine whether Eribulin Mesylate Administered in Combination with Pemetrexed is safe and tolerable and to gain a preliminary indication of clinical benefit when administered to Patients with Stage IIIB or IV Nonsquamous Non Small Cell Lung Cancer.

DETAILED DESCRIPTION:
This open-label, multicenter, randomized study will consist of a Phase Ib portion: a safety run-in period with 3 ascending doses of eribulin; and a Phase II portion: a randomized 3-arm design. .

Phase Ib-Patients will be recruited into cohorts, into one of two parallel arms evaluating different eribulin dosing schedules (Arm 1: eribulin on Day 1; Arm 2: eribulin on Days 1 and 8), with a minimum of 3 and a maximum of 6 patients per cohort. All patients will receive pemetrexed (500 mg/m2) in combination with eribulin. All patients in a cohort will receive the same dose level of eribulin and there will not be any intra-patient dose escalation.

The dose level of eribulin will be escalated for additional cohorts in each of the two arms unless greater than or equal to 2 dose limiting toxicities (DLTs) are reported at the lower dose level(s) prior to enrollment of the next dose level.

Phase II- Patients will be randomized in a 1:1:1 ratio to receive either eribulin in combination with pemetrexed, in each of two dosing schedules (Arms 1 and 2), or pemetrexed alone (Arm 3). For both the Phase Ib and II portions, 1 cycle of therapy will last 21 days, with an estimated number of 6 cycles. Radiologic examinations including a computed tomography (CT) scan of the chest, abdomen, and pelvis as appropriate (and CT or magnetic resonance imaging [MRI] as appropriate), will be performed during Screening and thereafter every 2 cycles until disease progression.

ELIGIBILITY:
Inclusion Criteria:

Patients may be entered in the study only if they meet all of the following criteria:

1. Male or female patient greater than or equal to 18 years of age;
2. Histologically or cytologically confirmed nonsquamous NSCLC stage IIIB with malignant pleural effusion or stage IV disease not amenable to curative therapy. Patients with history of stage III disease that have relapsed after chemo- and radiotherapy are also eligible;
3. Have at least 1 site of measurable disease by the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST) criteria;
4. Have failed 1 prior platinum-doublet containing chemotherapy regimen for stage IIIB with malignant pleural effusion or stage IV nonsquamous NSCLC. One additional cytotoxic regimen is allowed for neoadjuvant, adjuvant, or neoadjuvant plus adjuvant therapy for Phase II patients. For patients enrolled in the Phase Ib portion, a maximum of three total prior regimens is allowed.

   Definition of a Chemotherapy Regimen: Any platinum-doublet containing chemotherapy, that may also include biological or targeted agents, and/or humanized antibodies, given concomitantly, sequentially, or both, is considered 1 regimen. If, due to toxicity, the dosing of 1 or more of the components must be reduced, or 1 or more of the components of the regimen must be omitted, or 1 of the components must be replaced with another similar drug, the changed version of the original regimen is not considered a new regimen. However, if a new component, dissimilar to any of the original components, is added to the regimen, the new combination is considered a new regimen. If the treatment is interrupted for surgery or radiotherapy, and then continues with an unchanged schedule and components, that treatment is considered as one regimen despite the interruption.
5. Life expectancy of greater than 3 months;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) less than 1;
7. Patients must have adequate renal function as evidenced by calculated creatinine clearance greater than 45 mL/min per the Cockcroft and Gault formula;
8. Patients receiving daily treatment with non-steroidal anti-inflammatory agents (NSAIDS) are eligible. Patients with creatinine clearance 45-79 ml/min must be able to interrupt NSAIDS 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of pemetrexed;
9. Patients must have adequate bone marrow function as evidenced by absolute neutrophil count (ANC) greater than 1.5 x 10^9/L, hemoglobin greater than 9.0 g/dL (a hemoglobin less than 9.0 g/dL at Screening is acceptable if it is corrected to greater than 9 g/dL by growth factor or transfusion prior to first dose), and platelet count greater than 100 x 10^9/L;
10. Patients must have adequate liver function as evidenced by bilirubin less than 1.5 times the upper limit of the normal range (ULN), and alkaline phosphatase, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than 3 x ULN (in the case of liver metastases, less than 5 x ULN). If there are bone metastases, liver-specific alkaline phosphatase may be separated from the total and used to assess liver function instead of total alkaline phosphatase;
11. Male or female patients of child-producing potential must agree to use double barrier contraception, oral contraceptives, or avoidance of pregnancy measures during the study and for 90 days after the last day of treatment;
12. Females of childbearing potential must have a negative serum pregnancy test;
13. Females may not be breastfeeding; and
14. Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

Patients may be entered in the study only if they meet all of the following criteria:

1. Prior treatment with pemetrexed, epothilone, ixabepilone, patupilone, halichondrin B or halichondrin B-like compounds;
2. Received chemotherapy, targeted therapy, radiotherapy, surgery, or immunotherapy within the 30 days prior to commencing study treatment or have not recovered from all treatment-related toxicities to Grade less than 1, except for alopecia;
3. History of other malignancies except: (1) adequately treated basal or squamous cell carcinoma of the skin; (2) curatively treated, a) in situ carcinoma of the uterine cervix, b) prostate cancer, or c) superficial bladder cancer; or (3) other curatively treated solid tumor with no evidence of disease for greater than 5 years;
4. Presence of brain metastases, unless the patient has received adequate treatment at least 4 weeks prior to randomization, and is stable, asymptomatic, and off steroids for at least 4 weeks prior to randomization;
5. Received treatment in another clinical study within the 30 days prior to commencing study treatment or patients who have not recovered from side effects of an investigational drug to Grade less than 1, except for alopecia;
6. Are currently receiving any other treatment, including palliative radiotherapy for the tumor aside from control of symptoms;
7. Common Toxicity Criteria (CTC) greater than Grade 3 peripheral neuropathy;
8. Require therapeutic doses of vitamin K antagonists;
9. Uncontrolled pleural effusions, ascites, or other third space fluid collections;
10. Uncontrolled diabetes mellitus Type 1 or 2; Significant cardiovascular impairment (history of congestive heart failure greater than New York Heart Association (NYHA) Grade II, unstable angina or myocardial infarction within the past 6 months, or serious cardiac arrhythmia);
11. Patients with organ allografts requiring immunosuppression;
12. Known positive human immunodeficiency virus (HIV), known hepatitis B surface antigen, or hepatitis C positive;
13. Hypersensitivity to halichondrin B and/or halichondrin B chemical derivative; or Have any medical condition that would interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2010-06-10 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2015-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harish Dave, Study Director — Quintiles, Inc.
Locations (17):
- United States (6):
  - Tucson, Arizona
  - Denver, Colorado
  - Fort Myers, Florida
  - Mount Holly, New Jersey
  - Nashville, Tennessee
  - Tacoma, Washington
- Prague, Czechia
- Germany (2):
  - Freiburg im Breisgau
  - Heidelberg
- Italy (2):
  - Milan
  - Rome
- Ukraine (6):
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Sumy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 23 investigative sites in the United States, Germany, Italy, Ukraine, and the Czech Republic from 10 June 2010 to 18 March 2015.
Pre-assignment Details: A total of 15 participants were enrolled and treated in Phase 1b portion of the study and 83 participants were enrolled of which 80 participants received study treatment in Phase 2 portion of the study.
Groups:
- Phase 1b, Arm 1 - Cohort 1: 0.9 mg/m^2 Eribulin Plus Pemetrexed: Participants received intravenous (IV) bolus of eribulin 0.9 milligram per square meter (mg/m^2) in combination with IV infused pemetrexed 500 mg/m^2 on Day 1 of each 21-day treatment cycle. Participants within the same cohort received the same dose of eribulin. Participants also received dexamethasone and vitamin supplements as recommended in the prescribing information for pemetrexed. The dose of eribulin was escalated to 1.4 mg/m^2 in Cohort 2 of Arm 1.
- Phase 1b, Arm 1 - Cohort 2: 1.4 mg/m^2 Eribulin Plus Pemetrexed: Participants received IV bolus of eribulin 1.4 mg/m^2 in combination with IV infused pemetrexed (500 mg/m^2) on Day 1 of each 21-day treatment cycle. Participants within the same cohort received the same dose of eribulin. Participants also received dexamethasone and vitamin supplements as recommended in the prescribing information for pemetrexed. The dose of eribulin was not further escalated.
- Phase 1b, Arm 2 - Cohort 1: 0.7 mg/m^2 Eribulin Plus Pemetrexed: Participants received IV bolus of eribulin 0.7 mg/m^2 on Days 1 and 8 of each 21-day treatment cycle. On Day 1 only of each 21-day treatment cycle, participants also received IV infused pemetrexed (500 mg/m^2). Participants within the same cohort received the same dose of eribulin. Participants also received dexamethasone and vitamin supplements as recommended in the prescribing information for pemetrexed. The dose of eribulin was not further escalated.
- Phase 2, Arm 1: 0.9 mg/m^2 Eribulin Plus 500 mg/m^2 Pemetrexed: Participants received IV bolus of eribulin 0.9 mg/m^2 in combination with IV infused pemetrexed (500 mg/m^2) on Day 1 of each 21-day treatment cycle. Dexamethasone and vitamin supplements were administered as recommended in the prescribing information for pemetrexed.
- Phase 2, Arm 2: 500 mg/m^2 Pemetrexed: Participant received IV infused pemetrexed (500 mg/m^2) alone on Day 1 of each 21-day treatment cycle. Dexamethasone and vitamin supplements were administered as recommended in the prescribing information for pemetrexed.
Period: Overall Study
Arm/Group | Phase 1b, Arm 1 - Cohort 1: 0.9 mg/m^2 Eribulin Plus Pemetrexed | Phase 1b, Arm 1 - Cohort 2: 1.4 mg/m^2 Eribulin Plus Pemetrexed | Phase 1b, Arm 2 - Cohort 1: 0.7 mg/m^2 Eribulin Plus Pemetrexed | Phase 2, Arm 1: 0.9 mg/m^2 Eribulin Plus 500 mg/m^2 Pemetrexed | Phase 2, Arm 2: 500 mg/m^2 Pemetrexed
Started | 4 | 6 | 5 | 42 | 41
Safety Population | 4 | 6 | 5 | 41 | 39
Modified Intent-to-treat (MITT) | 4 | 6 | 5 | 39 | 39
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 6 | 5 | 42 | 41
Not completed — Death | 2 | 2 | 1 | 19 | 19
Not completed — Completed 1 Year Follow-Up Per Protocol | 0 | 0 | 0 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1
Not completed — Administrative reasons | 0 | 0 | 0 | 0 | 1
Not completed — Progressive disease | 0 | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1
Not completed — Other | 2 | 4 | 4 | 16 | 15

BASELINE CHARACTERISTICS:
Population: All Enrolled Participants.
Groups:
- Phase 1b, Arm 1 - Cohort 1: 0.9 mg/m^2 Eribulin Plus Pemetrexed: Participants received IV bolus of eribulin 0.9 mg/m^2 in combination with IV infused pemetrexed 500 mg/m^2 on Day 1 of each 21-day treatment cycle. Participants within the same cohort received the same dose of eribulin. Participants also received dexamethasone and vitamin supplements as recommended in the prescribing information for pemetrexed. The dose of eribulin was escalated to 1.4 mg/m^2 in Cohort 2 of Arm 1.
- Total: Total of all reporting groups
Arm/Group | Phase 1b, Arm 1 - Cohort 1: 0.9 mg/m^2 Eribulin Plus Pemetrexed | Phase 1b, Arm 1 - Cohort 2: 1.4 mg/m^2 Eribulin Plus Pemetrexed | Phase 1b, Arm 2 - Cohort 1: 0.7 mg/m^2 Eribulin Plus Pemetrexed | Phase 2, Arm 1: 0.9 mg/m^2 Eribulin Plus 500 mg/m^2 Pemetrexed | Phase 2, Arm 2: 500 mg/m^2 Pemetrexed | Total
Number analyzed (Participants) | 4 | 6 | 5 | 42 | 41 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 6 | 5 | 29 | 27 | 69
  >=65 years | 2 | 0 | 0 | 13 | 14 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 16 | 14 | 34
  Male | 2 | 5 | 4 | 26 | 27 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 3 | 1 | 5
  Not Hispanic or Latino | 4 | 5 | 5 | 39 | 40 | 93
  Not reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-Limiting Toxicity (DLTs)
Description: DLT were defined as clinically significant adverse events (AE) occurring less than or equal to (<=) 21 days after treatment. Events as: Non-hematological: 1) Grade greater than or equal to (>=) 3 peripheral neuropathy; 2) Grade >=3 nausea, vomiting despite optimal antiemetic treatment; 3) Any nonhematologic toxicity of Grade >=3, with exceptions as alopecia, single laboratory values out of normal range, hypersensitivity reaction. Hematological:1) Grade 4 neutropenia lasting >7 days; 2) Febrile neutropenia as fever >=38.5 degree Celsius with absolute neutrophil count less than (<)1.0*10^9 per liter(/L); 3) Grade 3 thrombocytopenia with nontraumatic bleeding requiring platelet transfusion; 4) Grade 4 thrombocytopenia with/without nontraumatic bleeding. Other 1) Study drug related death; 2) Toxicity that dose escalation committee believed to be DLT that was not covered by above DLT criteria.
Time Frame: Cycle 1 (cycle length=21 days)
Population: Phase 1b Safety Analysis Set was defined as all participants enrolled into the Phase 1b portion of this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Arm 1 - Cohort 1: 0.9 mg/m^2 Eribulin Plus Pemetrexed | Phase 1b, Arm 1 - Cohort 2: 1.4 mg/m^2 Eribulin Plus Pemetrexed | Phase 1b, Arm 2 - Cohort 1: 0.7 mg/m^2 Eribulin Plus Pemetrexed
Number analyzed (Participants) | 4 | 6 | 5
Participants
  Alanine transaminase (ALT) increased (grade 3) | 0 | 1 | 1
  Aspartate transaminase (AST) increased (grade 3) | 0 | 1 | 0
  Febrile neutropenia (grade 4) | 0 | 1 | 0
  Neutropenia (grade 4) | 0 | 1 | 0
  Pneumonia (grade 4) | 0 | 0 | 1
  Thrombocytopenia (grade 4) | 0 | 1 | 0

2. Primary Outcome: Phase 1b: Percentage of Participants With Grade 3 or Higher Treatment Emergent Adverse Events (TEAEs)
Description: Safety assessment included monitoring and recording all AE including all Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 grades (for both increasing and decreasing severity), and serious adverse events (SAE); regular monitoring of hematology, blood chemistry, and urine values; periodic measurement of vital signs and electrocardiograms (ECGs); and performance of physical examinations. A TEAE was defined as an AE that had on onset date, or a worsening in severity from Baseline (pretreatment), on or after the first dose of study drug up to the end of the study. As per CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to AE.
Time Frame: From date of first dose up to 30 days after the last dose of study drug in Phase 1b, up to approximately 1 year 2 months
Population: Phase 1b Safety Analysis Set was defined as all participants enrolled into the Phase 1b portion of this study.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1b, Arm 1 - Cohort 1: 0.9 mg/m^2 Eribulin Plus Pemetrexed | Phase 1b, Arm 1 - Cohort 2: 1.4 mg/m^2 Eribulin Plus Pemetrexed | Phase 1b, Arm 2 - Cohort 1: 0.7 mg/m^2 Eribulin Plus Pemetrexed
Number analyzed (Participants) | 4 | 6 | 5
percentage of participants | 100.0 | 83.3 | 100.0

3. Primary Outcome: Phase 2: Percentage of Participants Who Experienced TEAEs
Description: Safety assessment included monitoring and recording all AE including all CTCAE version 4.0 grades (for both increasing and decreasing severity), and SAE; regular monitoring of hematology, blood chemistry, and urine values; periodic measurement of vital signs and ECGs; and performance of physical examinations. A TEAE was defined as an AE that had on onset date, or a worsening in severity from Baseline (pretreatment), on or after the first dose of study drug up to the end of the study.
Time Frame: From date of first dose up to 30 days after the last dose of study drug in Phase 2, up to approximately 3 years 6 months
Population: Phase 2 safety population included all participants enrolled and randomized to treatment in the Phase 2 portion of the study, except for those who (I) dropped out prior to receiving any study drug, (ii) were without any safety assessment following the first dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2, Arm 1: 0.9 mg/m^2 Eribulin Plus 500 mg/m^2 Pemetrexed | Phase 2, Arm 2: 500 mg/m^2 Pemetrexed
Number analyzed (Participants) | 41 | 39
percentage of participants | 97.6 | 94.9

4. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization until the earlier of the following two events: the date of progressive disease (PD) or the date of death. Progressive disease was defined as at least a 20 percent (%) increase in the sum of the longest diameter of target lesions (taking as reference the smallest sum on study), recorded since the treatment started or the appearance of 1 or more new lesions based on investigator assessments according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). If a participant did not progress, they were censored at the date of last tumor assessment, last known alive date, or until the start of a next line of therapy, whichever occurred first. PFS was estimated using Kaplan-Meier method and presented with 2-sided 95% confidence interval.
Time Frame: From the date of randomization until the earlier of the following two events: the date of PD or the date of death (Up to approximately 3 years 5 months)
Population: MITT population included all randomized participants who received at least one dose of study drug without major protocol eligibility violations.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2, Arm 1: 0.9 mg/m^2 Eribulin Plus 500 mg/m^2 Pemetrexed | Phase 2, Arm 2: 500 mg/m^2 Pemetrexed
Number analyzed (Participants) | 39 | 39
weeks | 18.1 [8.43 to 34.14] | 22.0 [12.14 to 29.00]

ADVERSE EVENTS:
Time Frame: Phase 1b: From date of first dose up to 30 days after the last dose of study drug in Phase 1b (up to approximately 1 years 2 months); Phase 2: From date of first dose up to 30 days after the last dose of study drug in Phase 2 (up to approximately 3 years 6 months)
Arm/Group | Phase 1b, Arm 1 - Cohort 1: 0.9 mg/m^2 Eribulin Plus Pemetrexed | Phase 1b, Arm 1 - Cohort 2: 1.4 mg/m^2 Eribulin Plus Pemetrexed | Phase 1b, Arm 2 - Cohort 1: 0.7 mg/m^2 Eribulin Plus Pemetrexed | Phase 2, Arm 1: 0.9 mg/m^2 Eribulin Plus 500 mg/m^2 Pemetrexed | Phase 2, Arm 2: 500 mg/m^2 Pemetrexed
All-Cause Mortality (participants affected / at risk) | 2/4 | 2/6 | 1/5 | 19/41 | 19/39
Serious Adverse Events (participants affected / at risk) | 4/4 | 3/6 | 4/5 | 13/41 | 7/39
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 5/5 | 40/41 | 37/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b, Arm 1 - Cohort 1: 0.9 mg/m^2 Eribulin Plus Pemetrexed (N=4) | Phase 1b, Arm 1 - Cohort 2: 1.4 mg/m^2 Eribulin Plus Pemetrexed (N=6) | Phase 1b, Arm 2 - Cohort 1: 0.7 mg/m^2 Eribulin Plus Pemetrexed (N=5) | Phase 2, Arm 1: 0.9 mg/m^2 Eribulin Plus 500 mg/m^2 Pemetrexed (N=41) | Phase 2, Arm 2: 500 mg/m^2 Pemetrexed (N=39)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Oesophageal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Mucosal Inflammation (General disorders) | 1 | 1 | 0 | 0 | 0
Multi-Organ Failure (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 1 | 1
Sepsis Syndrome (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Myasthenic Syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b, Arm 1 - Cohort 1: 0.9 mg/m^2 Eribulin Plus Pemetrexed (N=4) | Phase 1b, Arm 1 - Cohort 2: 1.4 mg/m^2 Eribulin Plus Pemetrexed (N=6) | Phase 1b, Arm 2 - Cohort 1: 0.7 mg/m^2 Eribulin Plus Pemetrexed (N=5) | Phase 2, Arm 1: 0.9 mg/m^2 Eribulin Plus 500 mg/m^2 Pemetrexed (N=41) | Phase 2, Arm 2: 500 mg/m^2 Pemetrexed (N=39)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 6 | 14
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 3 | 7
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 3 | 13 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 4
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 4
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 2
Conjunctivitis Allergic (Eye disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 5 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 10 | 6
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 3
Asthenia (General disorders) | 2 | 0 | 1 | 5 | 1
Chest Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 2 | 4
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 2 | 6 | 12
Mucosal Inflammation (General disorders) | 1 | 0 | 1 | 3 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 5 | 2
Seasonal Allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 4 | 0
Candidiasis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Eye Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes Simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 3 | 4
Oral Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Sepsis Syndrome (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 2 | 1 | 11 | 15
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 1 | 10 | 14
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 0 | 3 | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Breath Sounds Abnormal (Investigations) | 0 | 0 | 2 | 0 | 0
C-Reactive Protein Increased (Investigations) | 0 | 0 | 0 | 3 | 1
Creatinine Renal Clearance Decreased (Investigations) | 0 | 0 | 0 | 1 | 3
Platelet Count Decreased (Investigations) | 0 | 2 | 1 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 3 | 4
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 0 | 1 | 8 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2
Headache (Nervous system disorders) | 1 | 0 | 1 | 2 | 4
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 4 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 3 | 3
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 2
Hot Flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes